CLINICAL TRIAL: NCT06775535
Title: Assessment of Neuronal Activation Accuracy and Stimulation Sensation in Patients with Closed-loop Spinal Cord Stimulation (CL-SCS) Therapy
Brief Title: Neuronal Activation Accuracy in Closed-loop Spinal Cord Stimulation
Acronym: NAA
Status: Recruiting | Type: Observational
Sponsor: Karel Hanssens (Other)
Responsible Party: Sponsor-Investigator, Karel Hanssens, MD, AZ Delta
Organization: AZ Delta (Other)
Other Study IDs: 51773; CME AZ Delta (Other: 21083); Belgium registration number (Other: B1172021000026)
Record Dates: First submitted 2024-10-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Neuropathic Pain; Persistent Spinal Pain Syndrome Type 2
MeSH Terms: conditions — Chronic Pain; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ECAP-controlled, closed-loop SCS — Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude

SUMMARY:
Observational, prospective, single-center to assess neuronal activation accuracy and stimulation sensation in patients with closed-loop spinal cord stimulation therapy.

DETAILED DESCRIPTION:
The study follow patients with chronic pain who received an EvokeTM spinal cord stimulator. The main aim of this study is to evaluate what influence different settings on nerve activation have and how this affects patients' sensation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is deemed a suitable candidate for SCS trial and permanent implant and has been routinely scheduled to undergo an SCS trial phase with the Evoke SCS System.
* Subject has a minimum of pain intensity of 5/10 on the numeric rating scale (NRS) at baseline
* Subject is ≥ 18 years old.
* Subject is not pregnant or nursing.
* Subject is willing and capable of giving informed consent.

Exclusion Criteria:

* Subject currently has an active implantable device including pacemakers, spinal cord stimulator or intrathecal drug delivery system.
* Subject is incapable of understanding or responding to the study questionnaires.
* Subject is incapable of understanding or operating the patient programmer handset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from chronic pain and are eligible for SCS trial and permanent implant.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with change in stimulation sensation | 6-months
  Stimulation sensation will be characterized by study participants as better, worse or same for 5 different closed-loop sensitivity settings.

SECONDARY OUTCOMES:
NRS | Baseline, 3-months, 6-months, 12-months post-implant
  The numeric rating scale (NRS) is a pain screening tool. It is used to assess pain severity at that moment in time using a 0-10 scale. Zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Number of participants with reduced pain distribution | Baseline, 3-months, 6-months and 12-months post-implant
  Pain distribution will be assessed by showing a visual representation of the body that enables participants to indicate the locations of their pain.
Paraesthesia mapping | 3-months, 6-months and 12-months post-implant
  Paraesthesia mapping will be assessed by showing a visual representation of the body that enables participants to indicate the locations where they feel paraesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Hanssens, Principal Investigator — AZ Delta
Locations (1):
- AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No